CLINICAL TRIAL: NCT05723250
Title: Patient-Centered Video Education Intervention to Improve Rural Cancer Care Delivery in Vermont: a Feasibility Study
Brief Title: Care Coordination Educational Intervention Study for Patients from Rural Areas with Early Stage Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Randall F Holcombe, Director, UVM Cancer Center, University of Vermont Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 00002358
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: healthcare delivery; care coordination; early stage cancer; educational intervention
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Upfront Educational Intervention (Experimental): Participants will receive a video-based intervention after completing baseline survey instruments and prior to retesting after 4-6 months.
  Interventions: Other: Table-based Educational Intervention
- Delayed Educational Intervention (Experimental): Participants will complete baseline survey instruments and again complete surveys after 4-6 months. They will then receive the video-based educational tablet.
  Interventions: Other: Table-based Educational Intervention

INTERVENTIONS:
Other: Table-based Educational Intervention — Tablet based educational tool with videos about care coordination, cancer knowledge and self-advocacy.
  Other Names: Educational

SUMMARY:
Care Coordination is an essential component of cancer care delivery. Many patients experience poor care coordination. In this study, we hypothesize that provision of a video educational intervention to teach patients about cancer, care coordination and self-advocacy will improve patients' perception of care coordination. Cancer patients with early stage disease scheduled to receive adjuvant therapy, and who reside in a rural area, will be enrolled onto the study. Patients will be randomized to receive a table-based educational intervention tool initially (arm1) or after 4 months of therapy (arm2). Assessment of cancer knowledge, self-advocacy and care coordination will be obtained at baseline and after 4-6 months.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Breast, lung, or colon cancer diagnosis
* Stage I, II or III cancer
* Adjuvant chemotherapy started < 30 days or planned within the next 30 days
* Rural residence location in Vermont (outside Chittenden County)
* Proficient in English

Exclusion Criteria:

* History of prior malignancy treated with chemotherapy in last 3 years
* Known or suspected neuro-cognitive impairment
* Resident of Chittenden County, Vermont
* Patients with current diagnosis other than stage I, II or III breast, colon or lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Care Coordination Instrument Score | Baseline and 4 months
  Participants complete the Care Coordination Instrument (CCI), a 29-item questionnaire. Each item is rated on a Likert scale (Strongly Agree = 3 to Strongly Disagree = 0). A total score is generated by summing the item scores; possible total scores range from 0-87. Higher scores represent a greater perception of care coordination.

SECONDARY OUTCOMES:
Cancer Knowledge | Baseline and 4 months
  Participants complete the Cancer Knowledge Assessment Test (C-KAT). The test includes 5 multiple choice items. A total score is generated by summing the number of correct responses; total scores range from 0-5. Higher scores represent greater cancer knowledge.
Satisfaction with Educational Videos | 4 months
  Participants in the baseline intervention group complete the Satisfaction and Acceptability Questionnaire. This 5-item questionnaire assesses how helpful and easily accessible the educational videos were. There is also an open-ended question for other feedback. Answering yes to the items indicates greater satisfaction and ease of use.
Self-Advocacy Score | Baseline and 4 months
  Participants complete the Cancer Self-Advocacy Scale, a 20-item questionnaire. Each item is rated on a Likert scale (Strongly Agree = 6 to Strongly Disagree = 1). A total score is generated by summing the item scores; possible total scores range from 20-120. Higher scores represent greater self-advocacy skills.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Cancer Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request, with removal of PHI
Supporting Information: Study Protocol

REFERENCES:
- [Background] Okado I, Cassel K, Pagano I, Holcombe RF. Development and psychometric evaluation of a questionnaire to measure cancer patients' perception of care coordination. BMC Health Serv Res. 2020 Jan 21;20(1):52. doi: 10.1186/s12913-020-4905-4. PMID 31964391
- [Background] Okado I, Cassel K, Pagano I, Holcombe RF. Assessing Patients' Perceptions of Cancer Care Coordination in a Community-Based Setting. JCO Oncol Pract. 2020 Aug;16(8):e726-e733. doi: 10.1200/JOP.19.00509. Epub 2020 Mar 27. PMID 32216713
- [Background] Okado I, Pagano I, Cassel K, Holcombe RF. Perceptions of care coordination in cancer patient-family caregiver dyads. Support Care Cancer. 2021 May;29(5):2645-2652. doi: 10.1007/s00520-020-05764-8. Epub 2020 Sep 24. PMID 32970231